CLINICAL TRIAL: NCT05519553
Title: Peer Support Impact on Therapeutic Adherence in Patients With Multiple Sclerosis: a Mixed Methods Randomized Controlled Trial Pilot Study
Brief Title: Peer Support Impact on Therapeutic Adherence in Patients With Multiple Sclerosis
Acronym: PAIR-SEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC22_0175
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: multiple sclerosis; peer support; therapeutic adherence
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: a mixed methods randomized controlled trial
Masking Description: non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 30 MS (Multiple sclerosis, relapsing-remitting) patients
  Interventions: Other: Peer support
- Control group (No Intervention): 30 MS (Multiple sclerosis, relapsing-remitting) patients

INTERVENTIONS:
Other: Peer support — : 1 hour individual session with a peer support specialist at 1, 3 and 5 months after baseline
  Other Names: non applicable
  Arms: Experimental group

SUMMARY:
A mixed methods randomized controlled trial pilot study to assess peer support impact on relapsing-remitting multiple sclerosis patients' therapeutic adherence.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a debilitating and incurable chronic disease. Patients might benefit from peer support provided by patients entitled to give advice on daily life management with MS. Studies have shown that peer support can enhance chronic patients' quality of life in Psychiatry and Oncology.

This pilot study aims at assessing the impact of peer support on therapeutic adherence and quality of life in patients with MS, but also to appraise the project feasibility and acceptability among the healthcare team, with large-scale implementation in mind.

This mixed methods pilot study consists in a monocentric open-label randomized controlled trial. It is located in Nantes, France, and aims to recruit 60 patients with relapsing-remitting MS undergoing drug therapy from the Nantes University Hospital Neurology Department. Patients will be randomized 1:1 to receive either usual care only or usual care combined with peer support (3 individual sessions at 1, 3 and 5 months with a peer support specialist).

Primary outcome is enhanced therapeutic adherence 6 months after baseline, secondary outcomes include therapeutic compliance, quality of life, anxiety and depression, social support. All dimensions will be assessed using validated health questionnaires at baseline and at 6 months.

Interventions acceptability and feasibility will be evaluated using qualitative methods: undirected interviews with patients from the intervention group and 2 focus-groups, one with the peer support specialists and the other with the healthcare team.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* With relapsing-remitting MS according to 2017 revised Mc Donald criteria
* Attending medical consultation at Nantes University Hospital Neurology Department
* For whom background drug therapy is needed (oral or injectable)
* Who gave consent to participate in trial

Exclusion Criteria:

* Primary-progressive or secondary-progressive MS patients
* Patients under protection of vulnerable adults measure or convicted
* Patients not fluent in French
* Patients with severe cognitive impairment, who may find difficult filling out questionnaires properly
* Patients with a risk of follow-up interruption (move, nomadism…)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence | 6 months
  Description : score difference at baseline and 6 months of the " Necessity " and " Concerns " subscales of BMQ-Specific (Beliefs about medicines questionnaire) compared between control and intervention groups.
  A score, between 5 and 25, is calculated for each subscale by making a sum of the answers. Next, score difference between Necessity and Concerns (NCF) is calculated. NCF varies between -20 and +20. Value above 0 means that perceived treatment necessity exceeds treatment associated concerns. The more NCF comes close to +20, the better is the treatment risk/benefit balance.

SECONDARY OUTCOMES:
Therapeutic compliance | 6 months
  score difference at baseline and 6 months of MARS (Medication Adherence Rating Scale) questionnaire compared between control and intervention groups.
  A final score, between 5 and 25, is calculated by making a sum of the answers. If final score is 21 or above, or if every item is scored at least 4 points, the patient is deemed compliant.
Participants' quality of life | 6 months
  score difference at baseline and 6 months of MusiQoL-MCAT (Multidimensional Computerized Adaptive Short-Form Quality of Life Questionnaire Developed and Validated for Multiple Sclerosis) compared between control and intervention groups.
  The score on each dimension is obtained by computing the mean of the item scores for that dimension. All dimension scores are linearly transformed to a 0 to 100 scale. A global index score is computed as the mean of the dimension scores. Higher scores indicate a higher level of quality of life.
Emotional wellbeing | 6 months
  score difference at baseline and 6 months of HAD (Hospital Anxiety and Depression) questionnaire compared between control and intervention groups.
  A final score, between 0 and 21, is calculated by making a sum of the answers for each subscale. A subscale score >8 denotes anxiety or depression. The higher the score is, the worse the severity of depression or anxiety symptoms.
Social support | 6 months
  score difference at baseline and 6 months of SSQ6 (Social Support Questionnaire) compared between control and intervention groups.
  Two scores are calculated by making a sum of the answers in each dimension: N score (availability) ranges from 0 to 54 and S score (satisfaction) ranges from 6 to 36. Higher scores indicate a higher level of support availability or satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Leïla Moret, MD - PhD, Study Director — Nantes University Hospital; Sandrine Wiertlewski, MD, Principal Investigator — Nantes University Hospital

IPD SHARING:
Plan to Share IPD: No
non applicable

REFERENCES:
- [Derived] Guilmault L, Wiertlewski S, Malloggi L, Rousseau C, Jacq-Foucher M, Leclere B, Moret L. Peer support impact on therapeutic adherence in patients with multiple sclerosis: a mixed-methods pilot trial protocol. BMJ Open. 2023 Dec 30;13(12):e071336. doi: 10.1136/bmjopen-2022-071336. PMID 38159942